CLINICAL TRIAL: NCT03970928
Title: Comparison of Conventional Fluid Management With Pleth Variability Index Based Goal-directed Fluid Management in Elective Laparoscopic Hysterectomies.
Brief Title: Goal-directed Fluid Management Versus Conventional Fluid Management in Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gulseren Yilmaz, Principal Investigator, M.D., Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gulseren2
Record Dates: First submitted 2019-05-23; First posted 2019-06-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- goal-directed fluid management (GDFM) (Active Comparator): A pulse oximetry probe will be connected to the fourth finger of the hand in which there was not an arterial catheter in all patients and it will be wrapped so that it would not be affected by the external light. The pulse oximeter will then be connected to a monitor including the PVI software which automatically and continuously calculates the respiratory variations in the photoplethysmogram from data collected noninvasively via a pulse oximetry sensor. 0.9 % NaCl at a rate of 2 mL/kg/h will be infused in PVI- guided GDFM group, a 250-mL bolus crystalloid/colloid injection will be administered when PVI was higher than 13 % over 5 min.
  Interventions: Device: PVI
- Conventional fluid management group (CFMG) (No Intervention): This group will receive conventional fluid management described as follows: 0.9 % NaCl at a rate of 4- 8 mL/kg/h will be infused in CFGM group, a 250-ml bolus crystalloid/ colloid injection will be administered when the mean arterial blood pressure (MAP) decreased below 65 mmHg.

INTERVENTIONS:
Device: PVI — A pulse oximetry probe which transfers data to the monitor with software able to calculate PVI data. The monitor automatically and continuously calculates the respiratory variations in the photoplethysmogram from data collected noninvasively via a pulse oximetry sensor.
  Arms: goal-directed fluid management (GDFM)

SUMMARY:
Fluid management is critical in patients undergoing surgery. Goal-directed fluid management (GDFM) protocols have been shown to decrease the length of hospital stay. In this study, we aimed to compare the effects of conventional fluid management with Pleth Variability Index (PVI) guided on blood lactate, serum creatinine levels, postoperative kidney injury and the duration of hospital stay.

DETAILED DESCRIPTION:
Fluid management is critical in patients undergoing surgery. Goal-directed fluid management (GDFM) protocols have been shown to decrease the length of hospital stay in various kinds of surgical procedures. In this study, we aimed to compare the effects of conventional fluid management with Pleth Variability Index (PVI) guided on blood lactate, serum creatinine levels, postoperative kidney injury and the duration of hospital stay. Patients will be randomized to one of the study arms: group1 (conventional fluid management arm) will receive 0.9 % NaCl at a rate of 4- 8 mL/kg/h, a 250-ml bolus crystalloid/ colloid injection will be administered when the mean arterial blood pressure (MAP) decreased below 65 mmHg.; group 2 (GDFM); group 2 (GDFM group) will receive 0.9 % NaCl at rate of 2 mL/kg/h, a 250-mL bolus crystalloid/colloid injection will be administered when PVI is higher than 13 % over 5 min. In both groups, when MAP is still < 65 mmHg after fluid bolus infusion, 5 mg i.v. bolus ephedrine will be administered. The groups will be compared concerning postoperative blood lactate, serum creatinine levels, postoperative kidney injury and the duration of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Must be scheduled for laparoscopic hysterectomy Must be American Society of Anesthesiologists (ASA) class I-II-III

Exclusion Criteria:

- American Society of Anesthesiologists (ASA) class IV BMI > 40 kg/m2 Non-sinus heart rhythm MAP <65 mmHg at the onset of anesthesia induction Advanced renal and hepatic impairment Ejection fraction < 50 % Massive bleeding in the perioperative period

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
creatinine (mg/dl) | 3 hours after the operation
  Difference in serum creatinine levels between the two groups 3 hours after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Gulseren Yilmaz, MD, Principal Investigator — Kanuni Sultan Suleyman Hospital
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Please Enter the State Or Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No